CLINICAL TRIAL: NCT04105322
Title: Early Effects of Trunk Kinesio Taping on Balance and Functional Performance in Patients With Acute Stroke
Brief Title: Effects of Kinesio Taping on Balance and Functional Performance in Stroke Patients
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Banu BAYAR (Other)
Responsible Party: Sponsor-Investigator, Banu BAYAR, Prof Dr, Muğla Sıtkı Koçman University
Organization: Muğla Sıtkı Koçman University (Other)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 190135/133
Record Dates: First submitted 2019-09-23; First posted 2019-09-26 (Actual); Last update posted 2019-09-26 (Actual); Status verified 2019-09

CONDITIONS: Stroke, Acute; Hemiplegia; Balance; Functional Performance
Keywords: Acute stroke; Balance; Rehabilitation; Postural control
MeSH Terms: conditions — Stroke; Hemiplegia

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Kinesio Taping on Abdominal Muscles (Experimental)
  Interventions: Other: Kinesio Taping
- Kinesio Taping on Back Muscles (Experimental)
  Interventions: Other: Kinesio Taping
- Control (No Intervention)

INTERVENTIONS:
Other: Kinesio Taping — The kinesio tape is adhesive and it does not contain drug substance. After the patients were randomized to the groups, kinesio tape will be applied to the relevant region.
  Arms: Kinesio Taping on Abdominal Muscles; Kinesio Taping on Back Muscles

SUMMARY:
This study is planned to investigate the acute effects of trunk kinesio taping on balance and functional performance in acute stroke patients.

ELIGIBILITY:
Inclusion Criteria:

* 30-85 years
* Duration onset of stroke < 1 month Stroke time is between 0-1 months
* Score of Modified Rankin Scale 0-3
* Score of Mini Mental Test ≥ 24

Exclusion Criteria:

* Not volunteering to participate in the study
* Having another stroke history
* Having a history of fracture or surgical operation involving the lower extremity
* Have another neurological or orthopedic disorder affecting functionality
* Having visual or hearing problems
* Presence of skin lesions (decubitus ulcer, active infection, burns, malignancy, cellulite, scar, etc.) at the site of application.
* Allergic reaction to kinesio tape
* Being obese

Ages: 30 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 63 (Estimated)
Dates: Start 2019-09 (Estimated); Primary Completion 2020-03 (Estimated); Study Completion 2020-05 (Estimated)

PRIMARY OUTCOMES:
Trunk Impairment Scale | Change of trunk impairment from baseline at the end of 48 hours of each kinesio taping intervention.
  This scale comprises 17 items and evaluates static and dynamic sitting balance and trunk coordination. The items of the scale are scored on a 2-, 3- or 4-point ordinal scale. The total score ranges from a minimum of 0 to a maximum 23 points, higher scores indicate better performance.
Berg Balance Scale | Change of balance scores from baseline at the end of 48 hours of each kinesio taping intervention.
  The Berg balance scale is used to objectively determine a patient's ability (or inability) to safely balance during a series of predetermined tasks. It is a 14 item list with each item consisting of a five-point ordinal scale ranging from 0 to 4, with 0 indicating the lowest level of function and 4 the highest level of function.
Five Times Sit to Stand Test | Change of functional performance scores from baseline at the end of 48 hours of each kinesio taping intervention.
  This test reproduces the act of sitting and standing for five repetitions as rapidly as possible.
  The test performance was based on its duration; consequently, the shorter time taken by the patient, the better their functional condition would be.

SECONDARY OUTCOMES:
Wii Balance Board | Change of balance scores from baseline at the end of 48 hours of each kinesio taping intervention.
  The Basic Balance Test game will be used to assess the person's balance. At the end of this game is the routine evaluation of the device Wii Fit age; The patient's demographic characteristics, body mass index, weight transferred to the right and left foot and the Basic Balance Test will be calculated by the device using the game result. The fact that the resulting age is greater than the actual age of the patient will be considered as an inability to balance.
Postural Assessment Scale for Stroke | Change of postural ability from baseline at the end of 48 hours of each kinesio taping intervention.
  This scale contains 12 items for evaluating balance: 5 items to assess the maintenance of posture and 7 items to evaluate changes in posture. Each Postural Assessment Scale for Stroke item is rated on a scale from 0 to 3, for a maximum total score of 36: on this scale, the higher the score is, the more favourable the balance in stroke patients.
Patient Satisfaction: Visual Analogue Scale (VAS) | Change of patient satisfaction at the end of 48 hours of each kinesio taping application.
  It will be evaluated with the Visual Analogue Scale (VAS). The VAS consists of a 10 cm horizontal line. The left end of the line has the number 0 and the right end has the number 10. Number 0 means mad I'm not satisfied at all ken, while number 10 is considered "very satisfied". Satisfaction level increases from left to right on the line.

CONTACTS AND LOCATIONS:
Overall Officials: Asalet Aybüke GÜP, Bachelor, Principal Investigator — Muğla Sıtkı Koçman University; Banu BAYAR, Doctorate, Study Director — Muğla Sıtkı Koçman University

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Lee YJ, Kim JY, Kim SY, Kim KH. The effects of trunk kinesio taping on balance ability and gait function in stroke patients. J Phys Ther Sci. 2016 Aug;28(8):2385-8. doi: 10.1589/jpts.28.2385. Epub 2016 Aug 31. PMID 27630439
- [Background] Yazici G, Guclu-Gunduz A, Bayraktar D, Aksoy S, Nazliel B, Kilinc M, Yildirim SA, Irkec C. Does correcting position and increasing sensorial input of the foot and ankle with Kinesio Taping improve balance in stroke patients? NeuroRehabilitation. 2015;36(3):345-53. doi: 10.3233/NRE-151223. PMID 26409338
- [Background] Wang M, Pei ZW, Xiong BD, Meng XM, Chen XL, Liao WJ. Use of Kinesio taping in lower-extremity rehabilitation of post-stroke patients: A systematic review and meta-analysis. Complement Ther Clin Pract. 2019 May;35:22-32. doi: 10.1016/j.ctcp.2019.01.008. Epub 2019 Jan 17. PMID 31003662
- [Background] Rojhani-Shirazi Z, Amirian S, Meftahi N. Effects of Ankle Kinesio Taping on Postural Control in Stroke Patients. J Stroke Cerebrovasc Dis. 2015 Nov;24(11):2565-71. doi: 10.1016/j.jstrokecerebrovasdis.2015.07.008. Epub 2015 Aug 29. PMID 26321149
- [Background] Karatas M, Cetin N, Bayramoglu M, Dilek A. Trunk muscle strength in relation to balance and functional disability in unihemispheric stroke patients. Am J Phys Med Rehabil. 2004 Feb;83(2):81-7. doi: 10.1097/01.PHM.0000107486.99756.C7. PMID 14758293